CLINICAL TRIAL: NCT01000935
Title: Impact of Autologous Platelet Rich Plasma on Enhancing Repair of Rotator Cuff Tendons: A Multicentre Randomized Controlled Trial
Brief Title: Impact of Autologous Platelet Rich Plasma on Healing of Rotator Cuff Repairs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Dr. Helen Razmjou, Research Associate, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009-01
Record Dates: First submitted 2009-09-23; First posted 2009-10-23 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Rotator Cuff Pathology
Keywords: Rotator Cuff Decompression Repair

STUDY DESIGN:
Intervention Model Description: Intevention involved PRP injection
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma (Active Comparator): The platelet concentrate extracted from patient's own blood (PRP) will be applied to the surgical site after completion of the repair.
  Interventions: Other: Platelet Rich Plasma
- Surgical repair (standard-of-care) (No Intervention): Patients will have a rotator cuff repair without the PRP application.

INTERVENTIONS:
Other: Platelet Rich Plasma — Patient's blood will be drawn prior to the start of the procedure. The processing disposable (PD) size of 60ml will be used to yield 7 ml of Platelet concentrate volume. Using the lateral portal, the applicator for the PRP will be positioned in between the bone and the repaired rotator cuff without a cannula. The inflow will then be closed and the arthroscopic fluid will be aspirated via the outflow cannula. All other cannulae will be removed, producing a dry subacromial space. The PRP and autologous thrombin will then be transferred to the sterile field and drawn up into a dedicated spray applicator kit (Smartjet) and applied to the site of repair. A dry arthroscopic check will be performed to evaluate the clot formation of the applied solution.
  Arms: Platelet Rich Plasma

SUMMARY:
Partial-thickness and full-thickness rotator cuff tears are common soft-tissue conditions that often require surgical treatment. Initial efforts to improve tendon healing centered on improving the strength of the repair construct. More recent studies have focused on biologic enhancement of the healing process. The use of platelet concentrates to improve healing, has been explored considerably during the last decade. Platelet Rich Plasma (PRP) is a fraction of plasma that has been isolated and used to enhance regeneration in bone and soft tissues.

There is information on use of PRP in oral surgery, achilles tendon healing, limb lengthening procedures, chronic elbow tendinosis, ruptures/degenerative changes in the patellar tendon, and osteoarthritis of the knee. There are no randomized clinical trials to our knowledge that have examined the impact of PRP in patients with rotator cuff tear.

The objective of the proposed pilot study is to examine the effectiveness of autologous Platelet Rich Plasma (PRP) application in promoting healing of the rotator cuff (RC) tendons following arthroscopic rotator cuff repair through a randomized controlled study.

DETAILED DESCRIPTION:
Surgical procedures: Arthroscopic inspection of the shoulder will be performed to assess intra-articular structures and to evaluate the rotator cuff and other sub-acromial structures.

Arthroscopic Rotator Cuff Repair: Rotator cuff tears will be categorized as partial-thickness and full-thickness tears. The full-thickness tears will be classified as small (<1 cm), moderate (1-3 cm), and large (>3-5 cm) based on the largest dimension and will be treated with a repair using sutures and suture anchors as indicated.

Rehabilitation: A comprehensive protocol with instructions on different types of exercises will be provided pre-operatively. Rehabilitation will be based on the standard protocols for these procedures used at the Holland Centre.

Follow-ups: Patients will be monitored for 6 months, or when participation is terminated by the investigators, or because the patient withdrew consent or fails to return for visits. To evaluate safety, clinical laboratory (WBC, Hb, platelet count, serum chemistry and IL-6, CRP, PT, PTT and INR tests will be conducted at 6 weeks, and 3 months to determine the impact of treatment interventions.

ELIGIBILITY:
Inclusion criteria

1. Age >18 years
2. Diagnosis of partial or full-thickness rotator cuff tear of less or equal to 3 cm. confirmed by MRI or US within a period of 6 months prior to booking surgery.
3. The final inclusion will be based on arthroscopic assessment of the tear size and lack of significant concurrent pathology.

Exclusion Criteria

1. Unable to speak or read English
2. Non-repairable tear
3. Acute tears (<6 month)
4. Evidence of major joint trauma, infection, avascular necrosis, chronic dislocation, inflammatory arthropathy, frozen shoulder
5. Concurrent pathology of Superior Labral Anterior and Posterior (SLAP) lesions, Bankart lesions, or advanced osteoarthritis of the glenohumeral joint
6. Previous surgery of the affected shoulder
7. Bone marrow pathology
8. Abnormal platelet count
9. Serum hemoglobin concentration <11 g/dL or hematocrit <34%
10. Use of systemic cortisone
11. Current use of anticoagulants (i.e. Aspirin)
12. Use of an investigational drug and/or blood donation within the previous 3 months prior to surgery
13. Substance or alcohol abuse
14. Heavy smoking [a daily cigarettes consumption of more than 20 pieces, based on definition of the World Health Organization (WHO)]
15. Psychiatric illness that precludes informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-03; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Pain Scale | The primary outcome will be collected pre and post-operatively. The level of pain and medication utilization will be monitored throughout the study by completing a pain diary (day 1-30) and at 6 weeks, 3 months and 6 months following surgery.

SECONDARY OUTCOMES:
Adverse Effect | 6 months
Magnetic resonance Imaging (MRI) | 6 months after surgery
  The main secondary evaluation tool is the healing index examined by the post-operative MRI. In order to assess tendon healing, anatomic evaluation of the cuff repair will be done with use of a MRI as the investigation of choice. A postoperative MRI will be performed at a minimum of six months following surgery. The images will be reviewed by a senior radiologist who is blinded to patient group allocation.
Patient- focused outcomes | Before surgery and 3 and 6 months following surgery
  1. The SHORT Western Ontario Rotator Cuff Index
  2. The American Shoulder and Elbow Surgeons (ASES) form
  3. The Constant- Murley Score (CM) outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Richard Holtby, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holtby R, Christakis M, Maman E, MacDermid JC, Dwyer T, Athwal GS, Faber K, Theodoropoulos J, Woodhouse LJ, Razmjou H. Impact of Platelet-Rich Plasma on Arthroscopic Repair of Small- to Medium-Sized Rotator Cuff Tears: A Randomized Controlled Trial. Orthop J Sports Med. 2016 Sep 13;4(9):2325967116665595. doi: 10.1177/2325967116665595. eCollection 2016 Sep. PMID 27660800
- See also: Online access — http://journals.sagepub.com/doi/abs/10.1177/2325967116665595